CLINICAL TRIAL: NCT03103841
Title: Investigation of Sleep Quality and Prevalence of Sleep-disordered Breathing in Children and Young People With Epilepsy
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Collaborators: Action Medical Research (Other); University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: GN2392
Record Dates: First submitted 2016-12-12; First posted 2017-04-06 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2022-04

CONDITIONS: Epilepsy; Obstructive Sleep Apnea
Keywords: Children
MeSH Terms: conditions — Epilepsy; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children and young people with epilepsy: Sleep studies [Polysomnography] to assess presence and severity of obstructive sleep apnoea in children with epilepsy compared with a healthy control group
  Interventions: Procedure: Sleep studies [Polysomnography]
- Healthy controls: Sleep studies [Polysomnography] to assess presence and severity of obstructive sleep apnoea in children with epilepsy compared with a healthy control group
  Interventions: Procedure: Sleep studies [Polysomnography]

INTERVENTIONS:
Procedure: Sleep studies [Polysomnography] — Undertaking of sleep measurements by polysomnography and use of validated sleep questionnaires

SUMMARY:
Obstructive sleep apnoea (OSA) is a condition that affects around one in 20 children. In children with OSA, repeated episodes of airway obstruction can severely disturb and fragment sleep, leading to subsequent cognitive and behavioural problems .

Epilepsy affects 60,000 children in the UK and up to 30% of children with epilepsy have learning problems. Evidence suggests that OSA is more common in children with epilepsy, such that sleep disturbance could account for some of the learning problems they experience.

The aim of this study is to determine the prevalence of OSA in children with epilepsy. The investigators plan carry out detailed sleep studies in children with epilepsy and healthy controls to determine if children with epilepsy are more likely to have OSA than healthy children of the same age.

OSA is almost always treatable and the benefits of detecting and treating the condition in healthy children are well-established. If OSA proves to be a common finding in children with epilepsy, it will be important to carry out further studies to see if treating the condition has beneficial effects on learning and behaviour. This project could lead doctors to target sleep-disordered breathing as a way of improving learning outcomes in children with epilepsy.

DETAILED DESCRIPTION:
Obstructive sleep apnoea (OSA) is a condition that affects around one in 20 children. In OSA, the muscles and soft tissues in the throat relax and collapse during sleep causing the upper airway to become blocked. Breathing is briefly interrupted, blood oxygen levels fall and this causes the child to wake and start breathing again. These episodes can happen many times a night causing severely disturbed sleep. Untreated OSA may leave children with daytime attention difficulties and problems with learning and behaviour. Epilepsy affects approximately 60,000 children in the UK and up to 30 per cent of these children have associated learning problems.

There is evidence, including pilot work undertaken by the study team to suggest that OSA is more common in children with epilepsy, in which case, sleep disturbance could account for some of the learning problems they experience. The aim of this study is to determine the prevalence of OSA in children with epilepsy.

The investigators plan to carry out detailed polysomnography sleep studies in 55 children with epilepsy and 28 healthy children (controls). These studies will measure the length and quality of sleep over one night spent at the hospital. Seizure activity during this period will be monitored by video recordings combined with electroencephalograms (EEG). Sleep-disordered will be assessed using a variety of tests to measure air-flow, lung expansion and blood oxygen levels. This study should help to determine if children with epilepsy are more likely to have OSA than healthy children of the same age. OSA is almost always treatable and the benefits of detecting and treating the condition in healthy children are well-established.

If OSA proves to be a common finding in children with epilepsy, it will be important to carry out further studies to see if treating the condition has beneficial effects on learning and behaviour. This project could lead doctors to target sleep-disordered breathing as a way of improving learning outcomes in children with epilepsy.

Children with epilepsy attending Royal Hospital for Children, Edinburgh will be invited to take part in the study. Children without epilepsy (controls) will also be recruited. The children without epilepsy are included because although there are statistics for incidence of OSA in the general population, information for all the measures of sleep the team will collect are not available.

The study will assess sleep time, sleep efficiency, sleep architecture and respiratory events in children with epilepsy and control subjects.

To be sufficiently powered, it is planned to test 50 children with epilepsy and 25 healthy controls.

A sleep physiologist will work with participants to measure:

* Polysomnography (to record body functions in sleep - airflow in and out of the lungs, oxygen level in the blood, body position, breathing effort and rate, electrical activity of muscles, eye movement and heart rate)
* EEG or electroencephalography (to measure the electrical activity of the brain),
* Electrooculography (to measure rapid eye movements along horizontal and vertical axes),
* Chin electromyogram (to measure electrical impulses to chin muscles),
* Sleep quality.

A neurologist and physiologist will assess seizure frequency and discharges between seizures, and epilepsy types using video EEG monitoring. Further information will be collected: height, weight, body mass index, antiepileptic medication use, tonsillar size, Mallampati score (a measure of base of tongue to hard palate), completion of sleep questionnaires by participants and their parents, to include sleepiness scales and sleep quality index.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary epilepsy and attendance at Epilepsy clinic

Exclusion Criteria:

* Neurological co-morbidity affecting muscle tone OR any Respiratory co-morbidity including any history of asthma, airborne allergy or sleep-disordered breathing.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Apnea/Hypopnea index | Over study duration - 2 years
  Measurement of presence and severity of obstructive sleep apnoea

SECONDARY OUTCOMES:
Total Sleep Time | Over study duration - 2 years
  As measured on sleep study
Sleep Efficiency | Over study duration - 2 years
  Used to quantify sleep fragmentation i.e. %time asleep out of total study time
Sleep Quality | Up to 10 hours
  Pittsburgh Sleep Quality Index questionnaire
Symptoms of OSA | Over study duration - 2 years
  PSQ-SRBD scale questionnaire
Daytime Sleepiness | Over study duration - 2 years
  Epworth Sleepiness Score questionnaire

OTHER OUTCOMES:
Presence of epileptiform discharges during sleep | Single point in time measurement - Sleep study [8 to 10 hour period of sleep data]
  As measured on sleep EEG

CONTACTS AND LOCATIONS:
Overall Officials: Don S Urquhart, MD, FRCPCH, Principal Investigator — NHS Lothian
Locations (1):
- Royal Hospital for Sick Children, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Urquhart DS, Hill EA, Hill LE, Carruthers E, McLellan AE, Chin R, Shetty J. Adults with epilepsy appear to differ from children in regard to daytime sleepiness. J Clin Sleep Med. 2020 Aug 15;16(8):1393-1394. doi: 10.5664/jcsm.8528. PMID 32351204
- [Derived] Urquhart DS, McLellan AE, Hill LE, Carruthers E, Hill EA, Chin RF, Shetty J. A case-control study to investigate the prevalence of obstructive sleep apnea and the utility of the Sleep-Related Breathing Disorder scale of the Pediatric Sleep Questionnaire in children and young people with epilepsy. J Clin Sleep Med. 2024 Jul 1;20(7):1039-1047. doi: 10.5664/jcsm.11054. PMID 38318844